CLINICAL TRIAL: NCT05358561
Title: An Evaluation of the Effect of Grain-Like Products on Postprandial Glucose, Insulin and Subjective Saturation Response in Healthy Individuals
Brief Title: Postprandial Glucose, Insulin and Subjective Saturation Response in Healthy Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Özlem ÖZPAK AKKUŞ, Principal Investigator, Toros University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ChiaFlaxseed
Record Dates: First submitted 2022-04-22; First posted 2022-05-03 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Grain-Like Products; Postprandial Glucose; Plasma Insulin; Subjective Saturation Response; Healthy Individuals
Keywords: Carbohydrate; Chia; Flaxseed; Blood glucose; Insulin; Appetite
MeSH Terms: conditions — Insulin Resistance | interventions — Linseed Oil; Salvia hispanica seed extract

STUDY DESIGN:
Intervention Model Description: Cross over
Who Masked: Participant
Masking Description: Participants will not know what type of bread to eat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Nutritional analyzes applied to four cakes (No Intervention): The study is two-fold. In the preliminary study, the standard and test cakes (chia added cake, flax seed added cake, and chia+flax seed added cake) were developed and the amount of cake containing 50 g carbohydrate and the amount of moisture, ash, pulp, protein, fat, and digestible carbohydrate will be determined via analyses that will be carried at Toros University Food Chemistry Laboratory. Based on the results obtained, the amount of cakes containing 50 g digestible carbohydrate will be calculated and produced.
- Flaxseed cake (Experimental): Measuring blood glucose levels, plasma insulin and the satiety response levels of individuals after consumption of flaxseed cake
  Interventions: Dietary Supplement: Flaxseed and Chia
- Chia cake (Experimental): Measuring blood glucose levels, plasma insulin and the satiety response levels of individuals after consumption of chia cake
  Interventions: Dietary Supplement: Flaxseed and Chia
- Flaxseed and chia cake (Experimental): Measuring blood glucose levels, plasma insulin and the satiety response levels of individuals after consumption of flaxseed and chia cake
  Interventions: Dietary Supplement: Flaxseed and Chia
- Standart (Experimental): Measuring blood glucose levels, plasma insulin and the satiety response levels of individuals after consumption of standart cake
  Interventions: Dietary Supplement: Flaxseed and Chia

INTERVENTIONS:
Dietary Supplement: Flaxseed and Chia — Measuring blood glucose levels, plasma insulin and the satiety response levels of individuals after consumption of flaxseed, chia, flaxseed + chia and standart cakes
  Arms: Chia cake; Flaxseed and chia cake; Flaxseed cake; Standart

SUMMARY:
This study is a pioneering study in which the effect of the consumption of cakes produced with the addition of cereal-like products such as chia and flax seeds, which have high soluble fiber content, on blood glucose and insulin values, and the effect on the satiety response of individuals after consumption of cakes, will be a pioneer in many subjects.

As a result of the study, the relationships between the changes in the investigated parameters and the possible changes in these parameters will be revealed. The results obtained suggest that foods rich in soluble fiber such as chia and flaxseed and foods produced with the possible synergetic effect of chia and flaxseed are used in healthy and safe products suitable for our consumption habits, and that these products are both protective and protective against the development of complications such as obesity and type 2 diabetes, cardiovascular diseases. The investigators think that it may also play a role in preventing its progress.

DETAILED DESCRIPTION:
The present study aimed to compare the effect of the consumption of the cake supplemented with cereal-like produces, such as chia or flaxseed, which have high soluble fiber content, on postprondial blood glucose and insulin values. It also aimed to evaluate its effect of individuals' saturation response after consumption, and to develop cake recipes involving chia and flax seed. The study is two-fold. In the preliminary study, the standard and test cakes (chia added cake, flax seed added cake, and chia+flax seed added cake) were developed and the amount of cake containing 50 g carbohydrate and the amount of moisture, ash, pulp, protein, fat, and digestible carbohydrate will be determined via analyses that will be carried at Toros University Food Chemistry Laboratory. Based on the results obtained, the amount of cakes containing 50 g digestible carbohydrate will be calculated and produced. In the main study, the effect of standard and test cakes containing 50 g digestible carbohydrates on postprandial blood glucose, insulin, and subjective saturation response will be investigated. The study will be conducted with 14 volunteers aged between 19 and years 64, with no acute or chronic disease, having a Body Mass Index (BMI) of 18.5-24.9 kg/m2, and with a Beck Depression Scale of 8 or less. Those using prescription drugs and/or fiber supplements, pregnant or lactating women, those consuming excessive alcohol (> 2 drinks/day), women in menstrual period, those having allergic reaction to chia or flaxseed will not be included in the study. Before the individuals are included in the study, anthropometric measurements will be taken, Beck Depression Scale will be administered in order to evaluate the depression status, and individuals will be informed about the purpose and content of the study, and signed Informed Consent Form will be obtained from all participants. The individuals participating in the study will come to the research center once a week for four weeks to consume the cakes. Individuals will stay hungry for 10-12 hours after eating their usual dinner the night before the test and they will only consume water during this period. Baseline/fasting appetite responses of the individuals who came to the research center after this fasting period will be measured with a 100-mm visual analog scale (VAS) and baseline/fasting blood samples will be taken. The cakes will be consumed within 10 minutes and appetite responses will be measured using the 100-mm Visual Analog Scala (VAS) at 15, 30, 60, 90, 120, 180 minutes, and then venous blood samples will be taken by the nurse-in-charge. During this three-hour period, the participants will not be allowed to leave the research center, nor will they be allowed to consume any other food. Blood samples will be analyzed at the Forum Yaşam Hospital Biochemistry Laboratory. Glucose values will be analyzed by UV test analysis and insulin values will be analyzed by the chemical immunoassay method. The data obtained will be compared with the appropriate statistical methods and interpreted in the light of the literature.

ELIGIBILITY:
Inclusion Criteria:

* The study will be conducted with 14 volunteers
* Aged between 19 and years 64
* No acute or chronic disease
* Body Mass Index (BMI) of 18.5-24.9 kg/m2
* Beck Depression Scale of 8 or less.

Exclusion Criteria:

* Using prescription drugs and/or fiber supplements
* Pregnant or lactating women
* Consuming excessive alcohol (> 2 drinks/day)
* Women in menstrual period
* Having allergic reaction to chia or flaxseed

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-19 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Flax Seed Cake and Blood Glucose Parameters | One day
  Measurement of blood glucose parameters seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of flax seed cake.
Flax Seed Cake and Plasma Insulin Levels | One day
  Measurement of plasma insulin levels seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of flax seed cake.
Flax Seed Cake and Satiety Response Measurements | One day
  Measurement of the satiety response seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of flax seed cake.
Chia Cake and Blood Glucose Parameters | One day
  Measurement of blood glucose parameters seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of chia cake.
Chia Cake and Plasma Insulin Levels | One day
  Measurement of plasma insulin levels seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of chia cake.
Chia Cake and Satiety Response Measurements | One day
  Measurement of the satiety response seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of chia cake.
Flax Seed and Chia Cake and Blood Glucose Parameters | One day
  Measurement of blood glucose parameters seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of flax seed and chia cake.
Flax Seed and Chia Cake and Plasma Insulin Levels | One day
  Measurement of plasma insulin levels seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of flax seed and chia cake.
Flax Seed Cake and Satiety Response Measurements | One day
  Measurement of the satiety response seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of flax seed and chia cake.
Standart Cake and Blood Glucose Parameters | One day
  Measurement of blood glucose parameters seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of standart cake.
Standart Cake and Plasma Insulin Levels | One day
  Measurement of plasma insulin levels seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of standart cake.
Standart Cake and Satiety Response Measurements | One day
  Measurement of the satiety response seven times (0. minute, 15. minute, 30. minute, 60. minute, 90. minute, 120. minute, 180. minute) within three hours after consumption of standart cake.

OTHER OUTCOMES:
Nutritional analysis of flax seed, chia, flax seed + chia cake and standart cakes | Five days
  The study is two-fold. In the preliminary study, the standard and test cakes (chia added cake, flax seed added cake, and chia+flax seed added cake) were developed and the amount of cake containing 50 g carbohydrate and the amount of moisture, ash, pulp, protein, fat, and digestible carbohydrate will be determined via analyses that will be carried at Toros University Food Chemistry Laboratory. Based on the results obtained, the amount of cakes containing 50 g digestible carbohydrate will be calculated and produced.

CONTACTS AND LOCATIONS:
Locations (1):
- Özlem ÖZPAK AKKUŞ, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data can be shared with permission of principal investigator

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-12-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT05358561/SAP_000.pdf